CLINICAL TRIAL: NCT03157427
Title: Clinical Evaluation of the Performance of a Difluoroethane-based Cyto-selective Cryotherapy to Treat Dark Spots on the Hand in 30 Volunteers.
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryobeauty (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A00068-45
Record Dates: First submitted 2017-05-03; First posted 2017-05-17 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Solar Lentigo
Keywords: Solar Lentigo, Cryotherapy, Difluoroethane

STUDY DESIGN:
Intervention Model Description: Patients will be treated on the randomized hand, the other hand is the comparator/control.
  Comparison between the treated hand and the control hand will be performed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRYOBEAUTY MAINS (Experimental): Cryotherapy medical device designed to treat solar lentigo on the randomized hand.
  Interventions: Device: CRYOBEAUTY MAINS
- Control (No Intervention): The non randomized hand is not teated.

INTERVENTIONS:
Device: CRYOBEAUTY MAINS — CYOBEAUTY MAINS diffuses Difluoroethane gas to the skin. The administration of the cryogenic gas is temperature controlled, accurate and contactless (by means of a spray nozzle), in small quantity (<1g) and during a predetermined short duration (3 seconds)
  Arms: CRYOBEAUTY MAINS

SUMMARY:
This study evaluates the performance of "CRYOBEAUTY MAINS", a Cyto-selective Cryotherapy based on Difluoroethane as a treatment of Solar Lentigines in 30 volunteers. Only one application of "CRYOBEAUTY MAINS" in one hand (right or left hand according to the randomization code).

ELIGIBILITY:
Inclusion Criteria:

* Phototype II to IV
* Subjects having brown spots (solar lentigo) on both hands, diameter ≤ 6 mm (at least 1 spot per hand).
* Accepting not to expose themselves to the sun (or artificial UV) during the study.
* Affiliated to a health insurance scheme in accordance with the French law on research involving the human subjects
* Informed, having undergone a general medical examination attesting to his / her ability to participate in the study.
* Having given informed written consent for their participation in the study.

Non inclusion Criteria:

* Having carried out aesthetic care (exfoliants, scrubs or self-tanning, manicure, hand care, UV ...) in the month prior to the start of the study, on the hands.
* Having applied a depigmenting product in the month prior to the start of the study, on the hands.
* Having carried out aesthetic care at a dermatologist (laser, IPL, peeling, depigmenting creams, cryotherapy ...), on the hands, during the last 6 months.
* Presenting dermatosis, autoimmune disease, systemic, chronic or acute illness, or any other condition that may interfere with the treatment or influence the results of the study (diabetic, circulatory, cold allergic, Raynaud's syndrome ...)
* Any general or local treatment (dermocorticoids, corticosteroids, diuretics, etc.) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being in an exclusion period from a previous study
* Being unable to comply to the protocole.
* Having Received over 4,500 euros compensation for his / her participation in clinical trials in the previous 12 months, including participation in this study.
* Vulnerable: being unable to give or refuse consent.
* Protected by the law (guardianship, curatorship, safeguard of justice ...).
* Unable to write or read in French.
* Can not be contacted by telephone.
* For female subjects:

  * Pregnant woman (or wanting to be pregnant during the study) or during breastfeeding.
  * Female not willing to use contraceptives.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of CRYOBEAUTY MAINS's performance | 8 weeks
  Hexsel scoring:
  1. > Very significant clearance (about 90%); only minor evidence of hyper pigmentation remains
  2. > Significant improvement (about 75%); some evidence of hyper pigmentation remains
  3. > Intermediate between marked and slight improvement; about 50% improvement in the appearance of hyper pigmentation
  4. > Some improvement (about 25%); however, significant evidence of hyper pigmentation remains
  5. > Hyperpigmentation has not changed since baseline
  6. > Worse (hyperpigmentation is worse than at baseline)

SECONDARY OUTCOMES:
Evaluation of solar lentigines numbers | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  Counting by enumeration of spots
Evaluation of solar lentigines numbers | 4 weeks
  Counting by enumeration of spots
Evaluation of solar lentigines numbers | 8 weeks
  Counting by enumeration of spots
Evaluation of solar lentigines colors | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  Colors assessment: by using Mexameter® MX 18
Evaluation of solar lentigines colors | 4 weeks
  Colors assessment: by using Mexameter® MX 18
Evaluation of solar lentigines colors | 8 weeks
  Colors assessment: by using Mexameter® MX 18
Assessment of pain intensity | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  VAS
Complication and adverse events rate | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  Any complications or adverse events related or not to the treatment will be collected and evaluated.
Complication and adverse events rate | 4 weeks
  Any complications or adverse events related or not to the treatment will be collected and evaluated.
Complication and adverse events rate | 8 weeks
  Any complications or adverse events related or not to the treatment will be collected and evaluated.
Assessment of ergonomic and device's readiness | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  Ergonomic and device's readiness questionnaire : 6 QCM questions are given to the participants
Assessment of volunteers feeling (QoL) | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  MelasQoL (Melasma. Quality of Life Scale)
Assessment of volunteers feeling (QoL) | 4 weeks
  MelasQoL (Melasma. Quality of Life Scale)
Assessment of volunteers feeling (QoL) | 8 weeks
  MelasQoL (Melasma. Quality of Life Scale)
Evaluation of CRYOBEAUTY MAINS's performance | 0 week : same-day following the CRYOBEAUTY MAINS treatment
  Hexsel scoring:
  1. > Very significant clearance (about 90%); only minor evidence of hyper pigmentation remains
  2. > Significant improvement (about 75%); some evidence of hyper pigmentation remains
  3. > Intermediate between marked and slight improvement; about 50% improvement in the appearance of hyper pigmentation
  4. > Some improvement (about 25%); however, significant evidence of hyper pigmentation remains
  5. > Hyperpigmentation has not changed since baseline
  6. > Worse (hyperpigmentation is worse than at baseline)
Evaluation of CRYOBEAUTY MAINS's performance | 4 weeks
  Hexsel scoring:
  1. > Very significant clearance (about 90%); only minor evidence of hyper pigmentation remains
  2. > Significant improvement (about 75%); some evidence of hyper pigmentation remains
  3. > Intermediate between marked and slight improvement; about 50% improvement in the appearance of hyper pigmentation
  4. > Some improvement (about 25%); however, significant evidence of hyper pigmentation remains
  5. > Hyperpigmentation has not changed since baseline
  6. > Worse (hyperpigmentation is worse than at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — CPCAD Nice
Locations (1):
- Cpcad Nice Hôpital Archet 2, Nice, France

IPD SHARING:
Plan to Share IPD: No